CLINICAL TRIAL: NCT06504134
Title: Gastroesophageal Reflux Disease Diagnostic Trial
Acronym: GERDT
Status: Not yet recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Collaborators: West China Hospital (Other); Ruijin Hospital (Other); Tongji Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); The Second Affiliated Hospital of Baotou Medical College (Other)
Responsible Party: Principal Investigator, Luowei Wang, MD, Clinical Professor, Changhai Hospital
Other Study IDs: GERDT
Record Dates: First submitted 2024-07-04; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: the Novel Esophageal Cell Collection Device — Using the novel cell collection device and the deep learning method to collect and classify esophogeal cell to identify if the participants are GERD patients

SUMMARY:
Gastroesophageal reflux disease (GERD) is a very common condition in clinical practice. In China, GERD affects nearly 150 million patients, whose quality of life are seriously impacted. Currently, the diagnosis of GERD primarily depends on the results of 24h reflux monitoring. However, such examination is under a quite low acceptability. As a result, a large number of patients were not diagnosed timely and accurately, and serious social problems are induced, such as drug abuse of proton pump inhibitor. Our team has previously developed a novel device for esophageal cell enrichment and established an internationally pioneering method of cytological screening for esophageal cancer based on cutting-edge deep learning technology. This project aims to develop multiple deep learning algorithms and establish an innovative method for diagnosis of GRED, using the novel esophageal cell enrichment technology. The research includes: 1) constructing deep learning algorithms for automatic esophageal inflammatory cells recognition and classification; 2) mining and extracting the key features of esophageal squamous cells and inflammatory cells under physician-AI interaction; 3) establishing a prediction model for GERD by integrating digital features of squamous cells and inflammatory cells and building a cloud-based automatic diagnosis system; 4) investigating the immuno-infiltration atlas of GERD and its diagnostic value based on the enriched inflammatory cells. The ultimate goal is to solve current clinical problems and realize rapid, convenient, and accurate diagnosis of GERD.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years and ≤85 years, male or female;
2. A visit was made for symptoms such as persistent reflux, heartburn, bloating, early satiety, and belching;
3. Patients volunteered to participate in the clinical trial, signed an informed consent form, and were able to cooperate with clinical follow-up.

Exclusion Criteria:

1. History of esophageal surgery;
2. Presence of dysphagia, esophagogastric fundal varices, or esophageal stenosis;
3. Presence of coagulation disorders or taking anticoagulant or antiplatelet drugs;
4. Those with a life expectancy of less than 5 years;
5. Persons with mental anomalies who are incapable of behavioral autonomy;
6. Other conditions that, in the judgment of the physician, preclude participation in the trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population who underwent testing with the novel esophageal cell collection device due to related symptoms from June 2024 to December 2027
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 60 minutes
  sensitivity and specificity

IPD SHARING:
Plan to Share IPD: No